CLINICAL TRIAL: NCT01259973
Title: Phase I Clinical Trial. Study of the Impact of Pharmacogenetic Markers in Predicting the Appearance of Extrapyramidal Symptomatology After the Treatment With Typical vs. Atypical Antipsychotics, in Healthy Volunteers
Brief Title: Typical Versus Atypical Antipsychotics; Occupation of Striatal Receptors and the Appearance of Extrapyramidal Symptomatology, in Healthy Volunteers
Acronym: APSEP
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Fundacion Clinic per a la Recerca Biomédica (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); University of Barcelona (Other)
Responsible Party: Miquel Bernardo Arroyo (Principal Investigator and Leader of Hospital Clinic psychiatric department), Hospital Clinic of Barcelona
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: TRA-065; 2009-016519-40 (EudraCT Number); TRA-065 (Other Grant/Funding Number: Dirección General de Terapias Avanzadas y Trasplantes. Ministerio de Sanidad y Política Social)
Record Dates: First submitted 2010-12-13; First posted 2010-12-15 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2011-01

CONDITIONS: Pharmacogenetics; Healthy
Keywords: Pharmacogenetics; Antipsychotics; Extrapyramidal Symptoms
MeSH Terms: interventions — Risperidone; Haloperidol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Risperidone (Experimental)
  Interventions: Drug: Risperidone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Haloperidol (Experimental)
  Interventions: Drug: Haloperidol

INTERVENTIONS:
Drug: Risperidone — 1 single dose of 2.5mg masked in 250 mL of peach juice, for 1 day. Oral administration.
  Arms: Risperidone
Drug: Placebo — 1 single dose of 2.5mL physiological serum masked in 250 mL of peach juice, for 1 day. Oral administration.
  Arms: Placebo
Drug: Haloperidol — 1 single dose of 5mg masked in 250 mL of peach juice, for 1 day. Oral administration.
  Arms: Haloperidol

SUMMARY:
The purpose of this study is to determine in healthy volunteers treated with typical or atypical antipsychotics -AP-, the relationship between genetic polymorphisms in cytochrome genes CYP2D6 (*3, *4, *5, *6 and Nxn) and CYP3A5 (*3) with antipsychotic pharmacokinetics, occupancy of striatal dopaminergic receptors and the appearance of extrapyramidal symptomatology -EPS-.

DETAILED DESCRIPTION:
Objective:

The preliminary results indicate that pharmacological factors (AP, dose and drug availability depending on cytochrome activity) are risk factors for AP-induced EPS.

In this clinical trial, the investigators will study, in healthy volunteers, the effects on pharmacokinetics, occupancy of striatal dopaminergic receptors and the appearance of EPS according to genetic polymorphisms in cytochrome genes CYP2D6 (*3, *4, *5, *6 and Nxn) and CYP3A5 (*3). The investigators will compare a typical AP (Haloperidol) with an atypical AP (Risperidone), both of which are metabolized by CYP2D6 and CYP3A5.

Specific objectives:

* Study the relationship between genetic polymorphisms in cytochrome genes CYP2D6 (*3, *4, *5, *6 and Nxn) and CYP3A5 (*3) and plasmatic levels of Haloperidol and Risperidone.
* Study the relationship between genetic polymorphisms in cytochrome genes CYP2D6 (*3, *4, *5, *6 and Nxn) and CYP3A5 (*3) and the grade of occupancy of striatal dopaminergic receptors with Haloperidol and Risperidone.
* Study the relationship between plasmatic levels of Haloperidol and Risperidone and the grade of occupancy of striatal dopaminergic receptors with these two drugs.
* Study the relationship between genetic polymorphisms in cytochrome genes CYP2D6 (*3, *4, *5, *6 and Nxn) and CYP3A5 (*3), plasmatic levels of Haloperidol and Risperidone, and the grade of occupancy of striatal dopaminergic receptors with these two drugs, with the appearance of AP-induced EPS.

Methodology:

From a cohort of 200 healthy volunteers (males and females with ages between 18-30 years), previously genotyped for CYP2D6 and CYP3A5 genes (from January to June 2010), the investigators have selected subjects depending on their metabolizer phenotype (poor metabolizers, intermediate metabolizers, extensive metabolizers and ultrarapid metabolizers) by DNA extraction from whole blood samples and SNP detection approaches.

Finally, the investigators will include the following four phenotypical groups with 6-8 subjects in each of the groups (a total of N=32 subjects, approximately):

* poor metabolizers (PM) CYP2D6*
* poor metabolizers (PM) CYP3A5**
* extensive metabolizers (EM) CYP2D6/CYP3A
* ultrarapid metabolizers (UM) CYP2D6*

The design corresponds to a three ways cross-over randomized and double-blind trial, with a wash-out period of one week among each treatment.

Measurements of occupancy of striatal dopaminergic receptors will be done by single photon emission computed tomography -SPECT- and SEP will be measured based on the Simpson-Angus scale and actimetry.

General protocol:

One week before their participation in the trial, volunteers will undergo clinical and physical explorations (blood test, electrocardiography, urine drug screening...) and will be trained in the different tests of the study (to minimize differences regarding to experience).

During the study, participants will be treated with a single dose of an AP drug (5mg Haloperidol or 2.5mg Risperidone) or a single dose of placebo (2.5mL physiological serum).

Plasma levels will be measured at +0.5h, +1h, +2h, +4h, +6h, +8h and +12h of drug/placebo administration.

The tracer [123I]IBZM will be administered at +3h of drug/placebo administration and SPECT will be performed at +5h.

Status of EPS, as well as positive and negative AP-derived symptoms, will be measured at -1h and at different time frames post-drug/placebo administration, beginning at +3h and until +24h (depending on each Scale used).

Participants will be hospitalized for three complete days (separated between them by one wash-out week after each treatment) from 8.00h to 8.00h of the following day at Phase I Unit of "Hospital de Sant Pau i de la Santa Creu", in Barcelona, in order to monitor the results obtained after each treatment. During their hospitalization, participants will be given food and drink every two hours.

This clinical trial will start in February 2011 and finish in November 2011.

ELIGIBILITY:
Inclusion Criteria that chosen participants must fulfill:

1. Subjects of both genders with ages between 18-30 years.
2. Subjects with normal values of clinical history and physical exploration.
3. Subjects without evidence of significant disease, organic or psychiatric, according to anamnesis (medical history), physical exploration and complementary tests.
4. Subjects with normal values of laboratory tests (hemogram and biochemical tests).
5. Subjects with normal values of vital signs (Blood pressure, Heart rate, Temperature) and Electrocardiography.
6. Female subjects must be using safe contraceptive methods, different from oral contraceptives.
7. Subjects could not have taken part in other clinical trials during the three previous months before to the beginning of this study.
8. Subjects could not have given blood during four weeks before the beginning of this study.
9. Subjects must accept freely their participation, with written informed consent.
10. After previous genotyping for CYP2D6 and CYP3A4/A5 genes, chosen participants must have one of the following genotypes of interest for this study:

    * poor metabolizers (PM) CYP2D6*
    * poor metabolizers (PM) CYP3A5**
    * extensive metabolizers (EM) CYP2D6/CYP3A
    * ultrarapid metabolizers (UM) CYP2D6*
11. Subjects must accept to undergo neuroimaging (SPECT).

Exclusion Criteria to reject potential participants:

1. Subjects with previous medical history of alcoholism or drug dependency.
2. Subjects with clinical history of allergy, idiosyncrasy or hypersensitivity to drugs.
3. Subjects with clinical history or current treatment with drugs whose metabolism could interfere in the action of CYP2D6 and CYP3A5 cytochromes, particularly if they are not able to give up the treatment for a period of 3-4 weeks before the beginning of the study and during its execution.
4. Subjects with clinical history or current consumption of drugs that could interfere in the action of CYP2D6 and CYP3A5 cytochromes (St John's wort, cruciferae, grapefruit ...), particularly if they are not able to give up their consumption for a period of 3-4 weeks before the beginning of the study and during its execution.
5. Subjects with contraindications for antipsychotic treatments due to: familiar/clinical history of hypersensitivity to antipsychotic drugs, deep depression of central nervous system, coma, Parkinson's disease.
6. Pregnant women, women in breastfeeding period or women that do not use safe contraceptive methods, different from oral contraception.
7. Subjects with positive serology for hepatitis B virus (HBV), hepatitis C virus (HCV) or human immunodeficiency virus (HIV).
8. Subjets with positive test in urine for ethanol, cannabis, cocaine, amphetamines, benzodiazepines and/or opiates.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-11 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Changes among genotypes in 24 h monitored Haloperidol and Risperidone pharmacokinetics | + 0.5h, +1h, +2h, +4h, +6h, +8h, +12h and +24h post-treatment
  Through a catheter, blood samples will be obtained at different time frames. Samples will be kept with anticoagulants and centrifuged immediately to separate the plasmatic fraction, which will be kept at -70ºC. In order to determine the concentration of Haloperidol (and reduced Haloperidol) and Risperidone (and 9-OH Risperidone), high performance liquid chromatography -HPLC- will be achieved.
  A poblation-pharmacokinetic model of the two AP drugs will be designed, and drug vs. placebo treatment results will be compared.
  Parameters determined: AUC, Cmax, Tmax, T(1/2), Vd, CL and MRT.
Changes from placebo in occupancy of striatal dopaminergic receptors by Haloperidol and Risperidone at 5h | +3h post-treatment: tracer injection. +5h post-treatment: image acquisition
  The tracer [123I]IBZM, a dopaminergic antagonist, will be administered by means of intravenous injection (at +3h post-treatment) at the opposite arm from which blood samples will be obtained. Neuroimaging will be done in SPECT gamma chambers and images will be quantified comparing drug vs. placebo treatment results.
  Parameters determined: Average Count Striatum and Count Occipital Cortex, Specific Uptake Ratio, D2 Occupational Receptor.
  100% of volunteers will undergo SPECT after placebo treatment and, among them, 50% after Haloperidol treatment and 50% after Risperidone treatment.
Changes from baseline in Extrapyramidal Symptomatology (EPS) at 3h, measured by Simpson-Angus Rating Scale (SARS)and Barnes Akathisia Rating Scale (BARS), and during 24 h, measured by actimetry | Heteroadministered scales will be measured at -1h pre-treatment (basal level) and at +3h. Actimetry will be measured continuosly since -1h pre-treatment until +24h
  AP-induced EPS measured by:
  * Heteroadministered scales:
    * Simpson-Angus Rating Scale (SARS). Assesses drug-induced parkinsonism (tremor, hypokinesia, rigidity, and postural instability).
    * Barnes Akathisia Rating Scale (BARS). Assesses drug-induced akathisia (restlessness and inability to sit still).
  * Actimetry: Continuous recording of movement, in terms of count of movements per minute, by using a wrist actimeter (model AW4) fitted to the arm not used for writing.
  Differences observed by comparing EPS after drug vs. placebo treatment will be considered.

SECONDARY OUTCOMES:
Changes from baseline in Positive and Negative Symptomatology at 3h, measured by Brief Psychiatric Rating Scale (BPRS) and Scale for the Assessment of Negative Symptoms (SANS), and at 24h, measured by Subjective Deficit Syndrome Scale (SDSS) | BPRS and SANS scales will be measured at -1h pre-treatment (basal level) and at +3h. SDSS scale will be measured at -1h pre-treatment (basal level) and at +24h
  AP-induced positive/negative symptoms measured by:
  * Brief Psychiatric Rating Scale (BPRS). Heteroadministered and semi structured interview (20 min) to determine hostility, suspiciousness, hallucination, and grandiosity.
  * Scale for the Assessment of Negative Symptoms (SANS). Heteroadministered interview (20 min) to determine affective blunting, alogia, avolition/apathy, anhedonia/asociality and disturbance of attention.
  * Subjective Deficit Syndrome Scale (SDSS). Autoadministered interview (20 min) to determine emotionless.
  Drug vs. placebo treatment will be compared.
Changes from baseline in 24h prolactin kinetics | At -1h pre-treatment (basal level) and at +0.5h, +1h, +2h, +4h, +6h, +8h, +12h and +24h post-treatment
  Blood samples analyzed will be the ones obtained for measuring plasmatic levels of antipsychotic drugs.
  Plasmatic levels of prolactin will be measured by enzymatic immunoassay approaches.
  Differences observed after drug vs. placebo treatment will be compared.
Changes from baseline in anticholinergic activity through Whole Saliva Test (WST) during 8h | At -1h pre-treatment (basal level) and at +1h, +2h, +4h, +6h and +8h post-treatment
  Salivette Containers (from Sarstedt) will be used to determine the saliva flow accumulated during 2 min.
  Differences observed after drug vs. placebo treatment will be compared.
Changes from baseline in cardiovascular effects through Orthostatism measurement during 8h | At -1h pre-treatment (basal level) and at +1h, +2h, +4h, +6h and +8h post-treatment
  In order to determine orthostatic hypotension, Systolic Arterial Pressure (SAP), Diastolic Arterial Pressure (DAP) and Cardiac frequency (CF) will be measured both after 3 min in supine position and after 3 min in erect position.
  Differences observed after drug vs. placebo treatment will be compared.
Changes from baseline in sedative effects during 8h | At -1h pre-treatment (basal level) and at +1h, +2h, +4h, +6h and +8h post-treatment
  AP-induced sedative effects measured by:
  * Psychomotricity
    * Flicker-Fusion Critical Frequency (FFCF). Detection of a flickering/stable red light.
    * Simple Reaction Time (SRT). Detection of a simple red light switched on/off.
    * Digit Symbol Substitution Test (DSST). Measures the amount of digits substituted correctly by its corresponding symbol.
    * Tapping Test (TT). Average of tappings per second.
  * Pupilometry. Detect pupil's response in basal conditions.
  * Visual Analog Scales (VAS). Detect agreement to a statement by indicating a position within two end-points.

CONTACTS AND LOCATIONS:
Overall Officials: Miquel Bernardo Arroyo, Head of Psychiatry, Principal Investigator — Hospital Clinic of Barcelona; Amalia Lafuente Flo, Pharmacology professor, Study Director — Dept. Pathologic Anatomy, Pharmacology and Microbiology, Medical Service, UB University of Barcelona; Sergi Mas Herrero, Pos-doc assistant professor, Study Chair — Dept. Pathologic Anatomy, Pharmacology and Microbiology, Medical Service, UB University of Barcelona; Patricia Gassó Astorga, Pos-doc associated professor, Study Chair — Dept. Pathologic Anatomy, Pharmacology and Microbiology, Medical Service, UB University of Barcelona; Gemma Trias Lafuente, Psychologist, Study Chair — Dept. Pathologic Anatomy, Pharmacology and Microbiology, Medical Service, UB University of Barcelona; Eva Ferrando Martorell, Pre-doc, Study Chair — Dept. Pathologic Anatomy, Pharmacology and Microbiology, Medical Service, UB University of Barcelona; Rosa M Antonijoan, Clinical Pharmacologist, Study Chair — Clinical Pharmacology Service, Hospital de la Santa Creu i Sant Pau; Analía Azaro, Clinical Pharmacologist, Study Chair — Clinical Pharmacology Service, Hospital de la Santa Creu i Sant Pau; Ignasi Carrió Gasset, Head of Nuclear Med Service, Study Chair — Nuclear Medicine Service, Hospital de la Santa Creu i Sant Pau; Manuel Barbanoj J Rodríguez, Head of Clinical Pharmacology, Head of Clinical Pharmacology, Study Chair — Clinical Pharmacology service, Hospital de la Santa Creu i Sant Pau
Locations (2):
- Spain (2):
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Clinic of Barcelona, Barcelona, Barcelona

REFERENCES:
- [Background] Lafuente A, Bernardo M, Mas S, Crescenti A, Aparici M, Gasso P, Catalan R, Mateos JJ, Lomena F, Parellada E. Dopamine transporter (DAT) genotype (VNTR) and phenotype in extrapyramidal symptoms induced by antipsychotics. Schizophr Res. 2007 Feb;90(1-3):115-22. doi: 10.1016/j.schres.2006.09.031. Epub 2006 Dec 5. PMID 17150335
- [Background] Lafuente A, Bernardo M, Mas S, Crescenti A, Aparici M, Gasso P, Deulofeu R, Mane A, Catalan R, Carne X. Polymorphism of dopamine D2 receptor (TaqIA, TaqIB, and-141C Ins/Del) and dopamine degradation enzyme (COMT G158A, A-278G) genes and extrapyramidal symptoms in patients with schizophrenia and bipolar disorders. Psychiatry Res. 2008 Nov 30;161(2):131-41. doi: 10.1016/j.psychres.2007.08.002. Epub 2008 Oct 15. PMID 18922583
- [Background] Crescenti A, Mas S, Gasso P, Parellada E, Bernardo M, Lafuente A. Cyp2d6*3, *4, *5 and *6 polymorphisms and antipsychotic-induced extrapyramidal side-effects in patients receiving antipsychotic therapy. Clin Exp Pharmacol Physiol. 2008 Jul;35(7):807-11. doi: 10.1111/j.1440-1681.2008.04918.x. Epub 2008 Mar 12. PMID 18346175
- [Background] Gasso P, Mas S, Bernardo M, Alvarez S, Parellada E, Lafuente A. A common variant in DRD3 gene is associated with risperidone-induced extrapyramidal symptoms. Pharmacogenomics J. 2009 Dec;9(6):404-10. doi: 10.1038/tpj.2009.26. Epub 2009 Jun 9. PMID 19506579
- [Background] Gasso P, Mas S, Crescenti A, Alvarez S, Parramon G, Garcia-Rizo C, Parellada E, Bernardo M, Lafuente A. Lack of association between antipsychotic-induced extrapyramidal symptoms and polymorphisms in dopamine metabolism and transport genes. Psychiatry Res. 2010 Jan 30;175(1-2):173-5. doi: 10.1016/j.psychres.2009.07.006. Epub 2009 Nov 5. PMID 19892410
- [Background] Ingelman-Sundberg M, Sim SC, Gomez A, Rodriguez-Antona C. Influence of cytochrome P450 polymorphisms on drug therapies: pharmacogenetic, pharmacoepigenetic and clinical aspects. Pharmacol Ther. 2007 Dec;116(3):496-526. doi: 10.1016/j.pharmthera.2007.09.004. Epub 2007 Oct 9. PMID 18001838
- [Background] Mauri MC, Volonteri LS, Colasanti A, Fiorentini A, De Gaspari IF, Bareggi SR. Clinical pharmacokinetics of atypical antipsychotics: a critical review of the relationship between plasma concentrations and clinical response. Clin Pharmacokinet. 2007;46(5):359-88. doi: 10.2165/00003088-200746050-00001. PMID 17465637
- [Background] Zanger UM, Turpeinen M, Klein K, Schwab M. Functional pharmacogenetics/genomics of human cytochromes P450 involved in drug biotransformation. Anal Bioanal Chem. 2008 Nov;392(6):1093-108. doi: 10.1007/s00216-008-2291-6. Epub 2008 Aug 10. PMID 18695978
- [Background] Catafau AM, Penengo MM, Nucci G, Bullich S, Corripio I, Parellada E, Garcia-Ribera C, Gomeni R, Merlo-Pich E; Barcelona Clinical Imaging in Psychiatry Group. Pharmacokinetics and time-course of D(2) receptor occupancy induced by atypical antipsychotics in stabilized schizophrenic patients. J Psychopharmacol. 2008 Nov;22(8):882-94. doi: 10.1177/0269881107083810. Epub 2008 Feb 28. PMID 18308793
- [Derived] Mas S, Gasso P, Fernandez de Bobadilla R, Arnaiz JA, Bernardo M, Lafuente A. Secondary nonmotor negative symptoms in healthy volunteers after single doses of haloperidol and risperidone: a double-blind, crossover, placebo-controlled trial. Hum Psychopharmacol. 2013 Nov;28(6):586-93. doi: 10.1002/hup.2350. Epub 2013 Oct 7. PMID 24519692